CLINICAL TRIAL: NCT02356679
Title: A Phase 4, Multicenter, Randomized, Open, Active Drug Comparative Trial to Evaluated the Efficacy and Safety of EUPASIDIN-S Tab. in Gastritis Patients
Brief Title: Efficacy and Safety of Eupasidin-s Tab.(EUPASIDIN-S) in Gastritis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EUPASIDIN-S_P4
Record Dates: First submitted 2014-09-02; First posted 2015-02-05 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2015-08

CONDITIONS: Acute Gastritis; Chronic Gastritis
MeSH Terms: interventions — DA 9601

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Eupasidin-s tab. (Experimental): three times per day, 1 tab for each time, PO, during 2weeks
  Interventions: Drug: Eupasidin-s Tab
- Stillen tab. (Active Comparator): three times per day, 1 tab for each time, PO, during 2weeks
  Interventions: Drug: Stillen Tab.

INTERVENTIONS:
Drug: Eupasidin-s Tab — three times per day, 1 tab for each time, PO, during 2weeks
  Other Names: Artemisia herb isopropanol soft ext. 60mg
  Arms: Eupasidin-s tab.
Drug: Stillen Tab. — three times per day, 1 tab for each time, PO, during 2weeks
  Other Names: Artemisia asiatica 95% ethanol ext. 60mg
  Arms: Stillen tab.

SUMMARY:
The purpose of this study is evaluate the Efficacy and Safety of EUPASIDIN-S Tab. in Gastritis Patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age is 19 years old and over, men or women
2. Patients diagnosed with acute or chronic gastritis by gastroscopy and need a treatment for gastritis symptoms
3. Patients with one or more erosions found by gastroscopy
4. Patients who voluntarily signed written informed consent may participate in the study

Exclusion Criteria:

1. Patients with peptic ulcer and gastroesophageal reflux disease
2. Patients with Gastrointestinal malignant tumor or surgery related to stomach resection
3. Patients with thromboembolism and coagulation disorder
4. Patients with significant cardiovascular, pulmonary, heptic, renal primary disease
5. Patients with abnormal laboratory result at screening

   * Aspartate aminotransferase(AST), Alanine aminotransferase(ALT), Creatinine > upper limit of normal range x 2
   * White blood cell(WBC) < 4,000/mm3
   * Platelet < 50,000/mm3
6. Patients administered with H2 receptor antagonists, proton pump inhibitors, muscarine receptor antagonists, other gastiritis treatment drug, protective factor builder, non-steroid anti-inflammatory drugs prior to study in 2 weeks
7. History of allergic reaction to the investigational product
8. Women either pregnant, breast feeding or possible to pregnant without contraceptive method
9. Use of other investigational drugs within 3 months prior to the study
10. Patients that investigators consider ineligible for this study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2014-08; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
cure rate of erosion | 2 weeks

SECONDARY OUTCOMES:
improvement rate of erosion | 2 weeks
improvement rate of erythema | 2 weeks
improvement rate of hemorrhage | 2 weeks
improvement rate of edema | 2 weeks
improvement rate of self symptoms | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sangyong Seol, Professor, Principal Investigator — Inje University Busanpaik Hospital
Locations (10):
- South Korea (10):
  - Inje University Busanpaik hospital, Busan, Busangjin
  - Chonbuk National University Hospital, Jeonju, Deokjin-gu
  - Chonnam National University Hospital, Guangju, Dong-gu
  - Wonju Severance Christian Hospital, Wŏnju, Ilsan-ro
  - Chungnam National University Hospital, Daejeon, Jung-gu
  - Wonkwang University School of Medicine & Hospital, Iksan, Muwang-ro
  - Yeungnam University Medical Center, Daegu, Nam-gu
  - Kosin University Gospel Hospital, Busan, Seo-gu
  - Dong-A University Hospital, Busan, Seo-gu
  - Hanyang University Medical Center, Seoul, Seongdong-gu